CLINICAL TRIAL: NCT00233051
Title: Expression of Inflammatory Mediators in Induced Sputum: A Potential Biomarker of Drug Response in COPD
Brief Title: Evaluating Genes in Sputum to Measure Drug Response in COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: E. Rand Sutherland, MD, MPH, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-1728
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Emphysema; Chronic Bronchitis
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Emphysema; Chronic Bronchitis; Inhaled Steroid; Salmeterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic | interventions — Fluticasone-Salmeterol Drug Combination

INTERVENTIONS:
Drug: Salmeterol or Salmeterol/Fluticasone

SUMMARY:
The purpose of this research study is to determine whether analysis of genes in sputum is a useful noninvasive technique for measuring response to drugs in patients with COPD.

We propose to use polymerase chain reaction to evaluate gene expression in induced sputum from adult current smokers with moderate COPD, adult former smokers with moderate COPD. This study is designed to determine whether changes in expression of previously-identified inflammatory markers in induced sputum can be detected in response to drug therapy in COPD and to evaluate potential differences in the expression of these markers in adult smokers with and without COPD. Pre- and post-treatment serum will be obtained to facilitate proteomic analysis of therapeutic response as well. Changes in sputum gene expression in response to treatment will be the primary outcome variable in this study. Secondary outcomes will include changes in lung function, as well as changes in induced sputum inflammation. These endpoints will be evaluated before and directly after 6 weeks of randomly-assigned treatment with either salmeterol xinafoate or fluticasone propionate/50mcg salmeterol xinafoate combination DPI bid. Endpoints will be re-evaluated following a 4 week wash-out period.

ELIGIBILITY:
Inclusion Criteria:

* Twenty adult subjects ≥ 40 years of age and ≥ 10 pack/year cigarette history will be evaluated.
* Subjects will be recruited such that one-half are current smokers and one-half are former smokers.
* All subjects will have COPD (FEV1/FVC < 70% and FEV1 => 40% predicted).
* Airway hyperresponsiveness and diffusion capacity for carbon monoxide will also be performed to more precisely characterize the physiologic phenotype in these subjects.

Exclusion Criteria:

* Subjects will be excluded if they have used inhaled or systemic corticosteroid or antibiotic use within 6 weeks or if they are currently treated with theophylline.
* A 6 weeks run off after an upper respiratory infection will be required for qualifying subjects.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Induced Sputum Gene Expression

SECONDARY OUTCOMES:
Lung Function

CONTACTS AND LOCATIONS:
Overall Officials: E Rand Sutherland, MD, MPH, Principal Investigator — National Jewish Medical and Research Center Faculty
Locations (1):
- National Jewish Medical and Research Center, Denver, Colorado, United States